CLINICAL TRIAL: NCT05025371
Title: The Role of Systemic Immuno-inflammatory Factors in Resectable Pancreatic Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Collaborators: Institutul Regional de Gastroenterologie & Hepatologie Prof. dr. Octavian Fodor (Other)
Responsible Party: Principal Investigator, Diana Schlanger, Dr., Iuliu Hatieganu University of Medicine and Pharmacy
Other Study IDs: SII-PDAC
Record Dates: First submitted 2021-08-26; First posted 2021-08-27 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-11

CONDITIONS: Pancreas Cancer, Duct Cell Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Systemic immune-inflammatory markers — Systemic immune-inflammatory markers used in this study: total neutrophil count, total lymphocyte count, total monocyte count, total platelet count, neutrophil-to-lymphocyte ratio (NLR), platelet-to-lymphocyte ratio (PLR), lymphocyte-to-monocyte ratio (LMR), systemic immune-inflammation index (SII), prognostic nutritional index (PNI)

SUMMARY:
Pancreatic cancer is a highly aggressive malignancy, its prognosis remaining poor despite the current advances in treatment. Systemic inflammatory reaction has been recently recognized as an important factor in the progression of cancer. The immune-inflammatory response has been measured through different scores or ratios, that combine the values of circulating immune cells, like neutrophil-to-lymphocyte ratio (NLR), platelet-to-lymphocyte ratio (PLR), lymphocyte-to-monocyte ratio (LMR), systemic immune-inflammation index (SII), prognostic nutritional index (PNI). The utility of these scores in different types of cancer has been more and more discussed. In pancreatic cancer, there has been no definite conclusion regarding the role of systemic immune-inflammatory factors; since controversies still exist, a deeper exploration of this subject, through more studies is welcomed. Our study intends to analyze the utility of systemic immune-inflammatory markers in resectable pancreatic cancer.

Our study is an observational cohort study, with retrospective data collection; it is a single-center study, that takes place in a hospital with experience in hepato-bilio-pancreatic surgery. The investigators intended to evaluate the role of the circulating immune cells (neutrophils, lymphocytes, monocytes) and different immune-inflammatory scores (NLR, LMR, PLR, SII, PNI) in predicting the overall survival of patients diagnosed with pancreatic ductal adenocarcinoma, that undergo curative surgical treatment. The investigators intended to assess the prognosis power of these factors in both preoperative and postoperative settings, as well as their dynamic after surgery. Through this study, the investigators hope to identify easy-to determine and easy-to-use markers that can be incorporated in clinical practice and that can effectively predict survival in pancreatic cancer patients. Nonetheless, the investigators want to explore the dynamic of the immune-inflammatory markers after curative surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pancreatic ductal adenocarcinoma
* Curative surgical procedure

Exclusion Criteria:

* Other histopathological types of pancreatic malignancies
* Palliative surgical interventions
* Incomplete/ insufficient data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated in the Surgical Department of Regional Institute of Gastroenterology and Hepatology Prof. Dr. O. Fodor Cluj-Napoca between January 2012 and December 2019
Sampling Method: Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | The last time of follow-up was April 2021

CONTACTS AND LOCATIONS:
Locations (1):
- Regional Institute of Gastroenterology and Hepatology "Prof. Dr. O. Fodor", Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schlanger D, Popa C, Pasca S, Seicean A, Al Hajjar N. The role of systemic immuno-inflammatory factors in resectable pancreatic adenocarcinoma: a cohort retrospective study. World J Surg Oncol. 2022 May 6;20(1):144. doi: 10.1186/s12957-022-02606-1. PMID 35513845